CLINICAL TRIAL: NCT04441957
Title: Endovenous MechanO-Chemical Ablation Plus Compression Versus CompreSSion Alone in Chronic Venous Ulcers Treatment
Brief Title: MechanO-Chemical Ablation Versus CompreSSion
Acronym: MOCASS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Belarusian State Medical University (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Vladimir Khryshchanovich, Professor, Belarusian State Medical University
Other Study IDs: 20140456
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Varicose Veins; Surgery
Keywords: VV; MOCA; GSV; Venous Ulcers
MeSH Terms: conditions — Varicose Veins; Varicose Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A, MOCA-group: Procedure/Surgery: MOCA Mechano-Chemical Ablation plus Elastic Compression
  Interventions: Device: Endovenous Mechano- Chemical Ablation
- Group B, Elastic Compression only group: Treatment: Elastic Compression only

INTERVENTIONS:
Device: Endovenous Mechano- Chemical Ablation — The Flebogrif™ catheter (Balton® Sp. z o.o., Warsaw, Poland) represents endoluminal Non Thermal Non Tumescent devices designed to cause occlusion (fibrosis) of the target vein through the combined mechanical and chemical damage to its endothelial lining with retractable cutters and foamed sclerosant.
  Other Names: MOCA
  Groups: Group A, MOCA-group

SUMMARY:
This study will be looking at the effect of Endovenous Mechano-Chemical Ablation (MOCA) in addition to multilayer elastic compression bandaging vs multilayer elastic compression bandaging only in patients with incompetent great saphenous vein (GSV) and venous ulcers (VU's).

DETAILED DESCRIPTION:
The most severe form of chronic venous disease is venous ulceration with an overall prevalence of about 1% in the adult population. Venous ulcers significantly impair quality of life, and their treatment places a heavy financial burden upon healthcare systems.

To get the ulcer to heal, the current best treatment is to wear a compression bandage with multiple layers, with which about 60% of these ulcers will heal within 6 months.

There is evidence that treatment of the varicose veins by sahenous veins stripping will prevent the ulcer recurrence.

Recent studies have suggested that novel proceduress of superficial truncal reflux elimination, such as foam sclerotherapy or treating the saphenous veins with termal (laser or radiofrequency) ablation to seal it effectively, may help the ulcers to heal more quickly and increase recurrence-free rate. These techniques can be carried out in the outpatient setting and are much better tolerated by patients in comparison to surgery.

At the same time, no studies which compared compression plus endovenous mechanochemical ablation (MOCA) vs. compression alone in chronic venous ulcers have been conducted to date.

The aim of this study is to see whether treatment of varicose veins using MOCA helps with healing.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age > 18 years.
2. Current leg ulceration of greater than 6 weeks.
3. Great saphenous vein (GSV) incompetence with reflux at least down to the knee level.
4. Primary symptomatic varicose veins, Clinical Etiological Anatomical Pathophysiological (CEAP) classification, clinical class C6.
5. Able to give informed consent to participate in the study after reading the patient information documentation.
6. Ankle Brachial Pressure Index (ABPI) ≥ 0.8.

Exclusion Criteria:

1. Postoperative varicose veins disease recurrence.
2. Patients who are unable to tolerate any multilayer compression bandaging / stockings will be excluded.
3. Deep venous thrombosis, thrombophilia associated with a high risk of deep venous thrombosis or postthrombotic syndrome.
4. History of pulmonary embolism or stroke.
5. Current anticoagulation therapy (within 7 days of enrollment).
6. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with GSV incompetence and C6 were included in in the prospective consecutive case study if they satisfied the selection criteria.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with varicose Veins from absent (score 0) to severe (score 3). | 6-12 months
  None (0), Few, scattered (1), Confined to calf or thigh (2) Involve calf and thigh (3)
Number of Participants with skin Pigmentation from absent (score 0) to severe (score 3). | 6-12 months
  None (0), Limited to perimalleolar area (1), Diffuse over lower third of calf (2), Wider distribution (above lower third of calf) (3)
Number of Participants with induration from absent (score 0) to severe (score 3). | 6-12 months
  None (0), Limited to perimalleolar area (1), Involving lower third of calf (2), Involving more than lower third of calf (3)
Number of Participants with active ulcers from absent (score 0) to severe (score 3). | 6-12 months
  None (0), 1 (1), 2 (2), more than 2 (3)
Number of Participants with active ulcer diameter from absent (score 0) to severe (score 3). | 6-12 months
  None (0), Diameter less than 2 cm (1), Diameter 2-6 cm (2), Diameter more than 6 cm (3)

SECONDARY OUTCOMES:
Number of Participants with ulcer recurrence-free rate (no - score 0, yes - score 1) | 3-24 months
  None (0), Less than 3 months (1), More than 3 months but less than 1 year (2) More than 1year (3)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir MD Khryshchanovich, Prof, Study Chair — Educational Institution "Belarusian State Medical University"
Locations (1):
- Educational Institution "Belarusian State Medical University", Minsk, Dzerzhinski Ave., 83,, Belarus

IPD SHARING:
Plan to Share IPD: Yes
To compare clinical efficacy of Endovenous Mechano-Chemical Ablation (MOCA) in addition to multilayer elastic compression bandaging and multilayer elastic compression bandaging only in patients with incompetent great saphenous vein (GSV) and venous ulcers (VU's).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12.2021
Access Criteria: To compare clinical efficacy of Endovenous Mechano-Chemical Ablation (MOCA) in addition to multilayer elastic compression bandaging and multilayer elastic compression bandaging only in patients with incompetent great saphenous vein (GSV) and venous ulcers (VU's).

REFERENCES:
- [Background] Kanchanabat B, Stapanavatr W, Kanchanasuttiruk P. Total superficial vein reflux eradication in the treatment of venous ulcer. World J Surg. 2015 May;39(5):1301-5. doi: 10.1007/s00268-014-2935-y. PMID 25680797
- [Background] Barwell JR, Davies CE, Deacon J, Harvey K, Minor J, Sassano A, Taylor M, Usher J, Wakely C, Earnshaw JJ, Heather BP, Mitchell DC, Whyman MR, Poskitt KR. Comparison of surgery and compression with compression alone in chronic venous ulceration (ESCHAR study): randomised controlled trial. Lancet. 2004 Jun 5;363(9424):1854-9. doi: 10.1016/S0140-6736(04)16353-8. PMID 15183623
- [Background] Gohel MS, Heatley F, Liu X, Bradbury A, Bulbulia R, Cullum N, Epstein DM, Nyamekye I, Poskitt KR, Renton S, Warwick J, Davies AH; EVRA Trial Investigators. A Randomized Trial of Early Endovenous Ablation in Venous Ulceration. N Engl J Med. 2018 May 31;378(22):2105-2114. doi: 10.1056/NEJMoa1801214. Epub 2018 Apr 24. PMID 29688123
- [Background] Sullivan LP, Quach G, Chapman T. Retrograde mechanico-chemical endovenous ablation of infrageniculate great saphenous vein for persistent venous stasis ulcers. Phlebology. 2014 Dec;29(10):654-7. doi: 10.1177/0268355513501301. Epub 2013 Aug 22. PMID 23969489
- [Background] Elias S, Raines JK. Mechanochemical tumescentless endovenous ablation: final results of the initial clinical trial. Phlebology. 2012 Mar;27(2):67-72. doi: 10.1258/phleb.2011.010100. Epub 2011 Jul 29. PMID 21803800